CLINICAL TRIAL: NCT04251806
Title: Sleep-disordered Breathing in Infants With Myelomeningocele
Status: Active, not recruiting | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, John Barks, Professor of Pediatrics, University of Michigan
Other Study IDs: HUM00165595; R01HL147261 (NIH)
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2024-12

CONDITIONS: Sleep-disordered Breathing; Myelomeningocele
Keywords: polysomnogram; development; sleep apnea
MeSH Terms: conditions — Sleep Apnea Syndromes; Meningomyelocele | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prenatal Repair: This group received prenatal myelomeningocele repair.
  Interventions: Diagnostic Test: neonatal polysomnography; Diagnostic Test: 2-year Bayley Exam; Diagnostic Test: 2-year polysomnography
- Postnatal Repair: This group received postnatal myelomeningocele repair.
  Interventions: Diagnostic Test: neonatal polysomnography; Diagnostic Test: 2-year Bayley Exam; Diagnostic Test: 2-year polysomnography

INTERVENTIONS:
Diagnostic Test: neonatal polysomnography — This procedure will allow the detection of sleep-disordered breathing in the neonatal period.
Diagnostic Test: 2-year Bayley Exam — This procedure will evaluate neurodevelopmental outcomes.
Diagnostic Test: 2-year polysomnography — This procedure will allow the detection of sleep-disordered breathing at 2 years of age.

SUMMARY:
This study aims to determine whether the risk for sleep-disordered breathing in infants with myelomeningocele (a severe form of spina bifida) differs among those who underwent fetal vs. postnatal surgery, and to examine the link between sleep-disordered breathing and neurodevelopment.

DETAILED DESCRIPTION:
Myelomeningocele (MMC), the most severe form of spina bifida, is characterized by exposure of the spinal cord through a spinal defect. Sleep-disordered breathing (SDB) is common in children with MMC and is a risk factor for sudden death. Abnormal sleep physiology is likely multifactorial, related to MMC level, brainstem dysfunction, musculoskeletal factors, and pulmonary abnormalities. In infants, SDB may be treatable with oxygen, caffeine, or positive airway pressure. Yet, SDB screening is not routine, even in centers with specialized MMC programs.

Evaluation of sleep in neonates who require intensive care is an emerging opportunity with potential for major impact on health and quality of life for affected children. As SDB and abnormal sleep are potentially treatable, early assessment and intervention could become an integral part of a multidisciplinary treatment strategy to optimize long-term medical and neurodevelopmental outcomes.

ELIGIBILITY:
Inclusion Criteria: neonates with myelomeningocele who are cared for at a study center NICU are eligible to participate after myelomeningocele repair.

Exclusion Criteria:

* born at <30 weeks gestation
* congenital anomalies that would predispose to sleep-disordered breathing (e.g. micrognathia)
* confirmed or suspected genetic syndromes that alter developmental outcomes

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Myelomeningocele is characterized by exposure of the spinal cord through a spinal defect.
Sampling Method: Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Evaluation of neonatal sleep-disordered breathing (SDB) in infants who had fetal versus postnatal myelomeningocele repair. | 35-42 weeks postmenstrual age
  Neonatal sleep studies will be used to capture neonatal Apnea-Hypopnea Index (AHI), the most widely accepted summary measure of sleep-disordered breathing severity for newborns who had fetal (prenatal) versus postnatal myelomeningocele repair.

SECONDARY OUTCOMES:
Association between neonatal sleep-disordered breathing and neurodevelopmental outcomes at 2 years of age for infants with myelomeningocele. | 22-26 months corrected age
  Bayley-IV developmental exams will be performed on all subjects around 2-years of age. The Bayley-IV will determine if the subject's level of thinking, language, and motor skills are similar to the level of most children their age. Our assessment will be based off the Cognitive Subscale Score. It has a range from 40-160 with a mean score of 100 and standard deviation of 15. The scores will analyzed with regression models and general linear models to see if there is an association between Neonatal AHI for infants with myelomeningocele, fetal vs. postnatal myelomeningocele repairs, and neurodevelopmental outcomes.
Persistence of sleep-disordered breathing at 2-years of age | 22-26 months corrected age
  Sleep studies will be performed at 2-years of age to capture AHI and compare to neonatal AHI for neonates who had fetal versus postnatal myelomeningocele repair.

CONTACTS AND LOCATIONS:
Overall Officials: John Barks, MD, Principal Investigator — University of Michigan
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Children's Hospital Colorado, Aurora, Colorado
  - Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Texas-Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://doi.org/10.1038/s41372-019-0468-9